CLINICAL TRIAL: NCT03001531
Title: Safety and Tolerance of Local Heat Application in the Paralyzed Area of Patients With Complete Paraplegia
Acronym: DecuHeat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-05
Record Dates: First submitted 2016-12-07; First posted 2016-12-23 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Perfusion; Complications
Keywords: Complete paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HydroSun (Active Comparator): application of ultraviolet light for 30 minutes
  Interventions: Device: HydroSun
- Hilotherm (Active Comparator): application of heat (maximum of 43°C) for 30 minutes
  Interventions: Device: Hilotherm

INTERVENTIONS:
Device: HydroSun — a skin area of the lower limb will be treated three times with ultraviolet light emitted by a halogen lamp
  Arms: HydroSun
Device: Hilotherm — a skin area of the lower limb will be treated three times with heat applied by a sleeve
  Arms: Hilotherm

SUMMARY:
Preconditioning of regional skin is known to reduce post surgery complications due to increased perfusion and better skin condition. The aim of this study is to prove that local heating through a standardized device in patients with spinal cord injury induces no burnings or other relevant side effects. The investigators expect an increased regional perfusion, temperature and redness.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* aged from 18 to 65 years
* paraplegia Th2-Th12
* spinal cord injury had occurred >12 weeks ago

Exclusion Criteria:

* infections
* fever
* diabetes
* heart failure stadium III
* renal insufficiency stadium III.
* scars, wounds or other injuries in the area of treatment
* skin type V and VI on Fitzpatrick scale

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
presence of burn injury | up to 24 hours
  grade 1 (hyperemia, redness), grade 2 a/b (blisters) and grade 3 (necrosis)

SECONDARY OUTCOMES:
blood perfusion | before and 1min after the application of light or heat
  perfusion (PeriFlux System 5000) in perfusion units
skin surface temperature | before and 1min after the application of light or heat
  measuring surface temperature with thermometer
skin redness | before and 1min after the application of light or heat
  visual inspection

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Switzerland

IPD SHARING:
Plan to Share IPD: No